CLINICAL TRIAL: NCT01064830
Title: A Single Center, Investigator-blinded Study of the Efficacy of Topical Cyclosporine 0.05% Ophthalmic Suspension (RESTASIS®) Under Occlusion Versus Vehicle in the Treatment of Brittle Nail Syndrome
Brief Title: Topical Cyclosporine Suspension for the Treatment of Brittle Nails
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, Aida Lugo-Somolinos, MD, Associate Professor, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 09-1141
Record Dates: First submitted 2010-02-05; First posted 2010-02-08 (Estimated); Results first posted 2012-12-03 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-02

CONDITIONS: Brittle Nail Syndrome
Keywords: brittle nail
MeSH Terms: conditions — Twenty-Nail Dystrophy | interventions — Cyclosporins

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- topical cyclosporine suspension (Active Comparator): apply 2 drops to 2 target nails under occlusion daily for 20 weeks
  Interventions: Drug: topical cyclosporine ophthalmic suspension 0.05%
- vehicle (Placebo Comparator): apply to target nails daily under occlusion daily for 20 weeks
  Interventions: Drug: vehicle

INTERVENTIONS:
Drug: topical cyclosporine ophthalmic suspension 0.05% — apply 2 drops to 2 target fingernails under occlusion daily
  Other Names: Restasis
  Arms: topical cyclosporine suspension
Drug: vehicle — apply 2 drops to 2 target fingernails under occlusion daily for 20 weeks
  Other Names: Refresh Dry Eye Therapy
  Arms: vehicle

SUMMARY:
Brittle nail syndrome (BNS) refers to nails that exhibit splitting, raggedness (fraying of the distal edge), and peeling (lamellar onychoschizia).(1) This is a common problem, affecting approximately 20% of women, with higher prevalence among the elderly.(2) A number of factors have been proposed as possible causes of nail brittleness, such as anemia, biotin deficiency, or cysteine deficiency. (3,4) However, most authors believe that brittle nails are usually caused by dehydration of the nail plate, either from repetitive cycles of hydration and dehydration related to hand washing or from exposure to dehydrating chemicals, such as those found in nail enamel and cuticle removers. (5,6) Inflammation of the nail as a potential contributing factor has never been studied.

There are currently not consistently effective treatments for this condition. Restasis® is effective in treating keratoconjunctivitis sicca. This condition is characterized by the troublesome condition of dry eyes partially due to decreased tear production exacerbated by inflammation. The BNS manifests itself by nail plate dehydration. The two conditions have in common disruption of water balance which gives rise to problematic clinical disorders. The hypothesis is that a product which benefits tear production would also be effective for brittle nails which contain roughly 15% water.

DETAILED DESCRIPTION:
Brittle nail syndrome (BNS) is a heterogeneous abnormality, characterized by increased fragility of the nail plate. About 20% of the population is affected by brittle nails and women are affected twice as frequently as men. (2). The diagnostic criteria for brittle nails are not well defined but most authors agree in at least these 3 criteria: onychoschizia (lamellar splitting of the free edge and distal portion of the nail plate), onychorrhexis (longitudinal thickening and thinning or ridging of the nail plate) and fraying or raggedness of the distal edge causing transverse splitting.

Although the cause of nail brittleness is unknown, most authors believe that it is caused by dehydration of the nail plate and that frequent cycles of hydration and dehydration as well as various mechanical and chemical insults increase the incidence of brittle nails. (7) The nail plate contains about 15% water and a very low lipid content so water permeation through the nail plate is high.(8) In fact, it has been demonstrated that the flux of water across the nail plate is 10 times more than the epidermis and 1000 times more permeable than the stratum corneum.(9) A recent report show that there was no significant difference in water content of brittle nails when compared to normal nails and suggested that nail plate water content is random and that nail plates are in a constant state of influx and efflux of water. (10) Keratoconjunctivitis sicca is a chronic, bilateral desiccation of the conjunctiva and cornea due to an inadequate tear film. There are two types: one caused by an inadequate tear volume and the other one caused by an accelerated tear evaporation due to poor tear quality (11). Restasis® (cyclosporine 0.05% topical emulsion) is effective in treating keratoconjunctivitis sicca.

BNS and keratoconjunctivitis sicca have in common a disruption of water balance which gives rise to problematic clinical disorders. We hypothesize that a product which improves corneal dehydration would also be effective for brittle nails. Our rationale for using occlusion is that is has been shown that occluding the skin with a vapor-permeable membrane increases the water flux and the barrier function is recovered at a normal rate. (12) We also hypothesize that using Restasis® (cyclosporine 0.05% topical emulsion) or its vehicle (Refresh Dry Eye Therapy®) under occlusion with a finger cot will increase the nail plate hydration balance and as a consequence will improve nail brittleness. Topical cyclosporine has been shown to be safe in the treatment of other dermatological conditions such as nail psoriasis and oral lichen planus. (13,14) An investigator-blinded design will differentiate if the observed effects are caused by the active ingredient in Restasis® (cyclosporine 0.05% topical emulsion) or its vehicle (Refresh Dry Eye Therapy®).

ELIGIBILITY:
Inclusion Criteria:

* • Must understand and voluntarily sign an informed consent form

  * Must be male or female and aged 18-75 years at time of consent
  * Must be able to adhere to the study visit schedule and other protocol requirements
  * At least 2 of the following: raggedness (fraying of the distal edge), splitting, and peeling (lamellar onychoschizia) of 2 target fingernails of the same hand. If the subject does not have 2 fingernails affected in the same hand, a second fingernail on the other hand may be used as control.
  * A direct microscopic examination with potassium hydroxide (KOH)/calcofluor that is negative for hyphae associated with dermatophytes
  * Women of childbearing potential must have a negative pregnancy test at enrollment

Exclusion Criteria:

* Inability to provide voluntary consent
* Pregnant or breastfeeding
* Fingernail fungal infection
* Use of any investigational medication within 4 weeks prior to start of study drug
* Subject has any known immunodeficiency or history of malignancy in the last 4 years, excluding nonmelanoma skin cancer.
* Use of any topical nail medication for 2 weeks
* Use of any topical nail product (nail polish, hardeners, acetone, etc) for 1 week prior to and during the study.
* Use of biotin 2 weeks before enrollment.
* No genetic nail abnormalities
* Known sensitivity to Restasis® or RDET®.
* Subject has psoriasis, lichen planus, or other abnormalities that could result in a clinically abnormal fingernail

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2010-02; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aida Lugo-Somolinos, MD, Principal Investigator — UNC- Chapel Hill
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Cyclosporine Solution 0.05% (Restasis®): Topical Cyclosporine 0.05% Ophthalmic Suspension
- Vehicle (Refresh Dry Eye Therapy®): Topical vehicle: Refresh Dry Eye Therapy® (ophthalmic solution of glycerin 1% and polysorbate 80 1%)
Period: Overall Study
Arm/Group | Cyclosporine Solution 0.05% (Restasis®) | Vehicle (Refresh Dry Eye Therapy®)
Started | 10 | 11
Completed | 8 | 7
Not Completed | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Cyclosporine Solution; Vehicle: apply to affected nails at night
- Total: Total of all reporting groups
Arm/Group | Cyclosporine Solution | Vehicle | Total
Number analyzed (Participants) | 10 | 11 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 10 | 18
  >=65 years | 2 | 1 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.0 (17.76) | 54.8 (10.02) | 51.6 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 11 | 19
  Male | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 10 | 11 | 21

OUTCOME MEASURES:

1. Primary Outcome: • Number of Patients Receiving at Least a 1-grade Improvement in the Physicians Global Improvement Assessment (PGIA) of Two Target Nails.
Description: IN a scale of 0-3 where 0 means normal nail and 3 means severe disease, the number of patients who received at least a decrease of 1 grade in the evaluation of two target nails
Time Frame: 20 weeks
Measure: Number; unit: patients
Groups:
- Cyclosporine Solution; Vehicle: topical
Arm/Group | Cyclosporine Solution | Vehicle
Number analyzed (Participants) | 10 | 11
patients | 10 | 11

2. Secondary Outcome: Patients Assessment of Satisfaction With Length of Fingernails
Description: the percentages of participants who were satisfied with the "length of fingernails"
Time Frame: 20 weeks
Population: all patients enrolled who completed this response measure at week 20.
Measure: Number; unit: percentage of patients
Groups:
- Cyclosporine Solution: cyclosporine solution
- Vehicle: vehicle
Arm/Group | Cyclosporine Solution | Vehicle
Number analyzed (Participants) | 9 | 8
percentage of patients | 44.4 | 12.5

ADVERSE EVENTS:
Arm/Group | Cyclosporine Solution | Vehicle
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 9/10 | 11/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cyclosporine Solution (N=10) | Vehicle (N=11)
upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
sinus infection (Infections and infestations) | 1 (1) | 1 (1)
ductal breast cancer (Stage 1 ) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
GI Virus (Gastrointestinal disorders) | 0 (0) | 1 (1)
herpes labialis (Infections and infestations) | 0 (0) | 1 (1)
influenza (Infections and infestations) | 1 (1) | 0 (0)
inner ear infection (Infections and infestations) | 0 (0) | 1 (1)
laryngitis (Infections and infestations) | 0 (0) | 1 (1)
poison ivy contact dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
rosacea (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
seasonal allergies (Immune system disorders) | 0 (0) | 1 (1)
sinusitis (Infections and infestations) | 1 (1) | 0 (0)
sinus congestion (Infections and infestations) | 0 (0) | 1 (1)
strept throat (Infections and infestations) | 1 (1) | 0 (0)
surgery for breast cancer (Reproductive system and breast disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No